

| Statistical and Epidemiological Analysis Plan | |
|---|---|
| BI Trial No.: | 1218.174 |
| Title: | Clinical characteristics, anti-hyperglycaemic treatment pattern and target attainment of type 2 diabetes mellitus patients in older population with or without albuminuria in China: A nationwide cross-sectional study |
| Responsible trial statistician: | Address: |
| | Phone: , Fax: |
| Responsible project epidemiologist: | |
| Date of statistical and epidemiological analysis plan: | 09Feb2018 |
| Version: | 1.0 |
| | Page 1 of 16 |
| | Proprietary confidential information International GmbH or one or more of its affiliated companies. All rights reserved. or in part - be passed on, reproduced, published or otherwise used without prior written permission. |

| Prepared by: | | |
|-------------------|--------------------|---|
| | 09 Feb 2018 | |
| Statistician | Date | |
| Approved by: | | |
| Approved by. | <b>a</b> 3 | |
| TrialStatistician | Date Date | |
| Clinical Projec | 09 Treb 2018 Date | |
| Project | Dage Feb nows | _ |

# **TABLE OF CONTENTS**

| TA | BLE ( | OF CONTENTS | 3 |
|---|---|---|---|
| 1. | $\mathbf{L}$ | IST OF ABBREVIATIONS | 4 |
| 2. | | NTRODUCTION | |
| 3. | | HANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. ( | | OMES | |
| | .1 | MAIN OUTCOMES | |
| | | | 7 |
| | .3 | OTHER VARIABLES | |
| 6. ( | GENE: | RAL ANALYSIS DEFINITIONS | 8 |
| 6 | .1 | EXPOSURE | |
| 6 | .2 | IMPORTANT PROTOCOL VIOLATIONS | |
| 6 | .3 | PATIENT SETS ANALYSED | |
| | | | 8 |
| _ | .5 | HANDLING OF MISSING DATA AND OUTLIERS | |
| | .6 | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | | LANNED ANALYSIS | |
| | .1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| | .2 | CONCOMITANT DISEASES AND MEDICATION | |
| | .3 | METHODS ADDRESSING BIAS | 11 |
| 7 | .4 | METHODS ADDRESSING CONFOUNDING / EFFECT MEASURE | |
| _ | | MODIFICATION | |
| 7 | .6 | MAIN ANALYSES | 11<br>11 |
| 7 | .8 | EXPOSURE TIME | |
| | .0<br>.9 | SAFETY ANALYSIS | |
| , | 7.9.1 | Adverse events | |
| | 7.9.2 | Laboratory data | |
| | 7.9.3 | Vital signs | |
| | 7.9.4 | ECG | |
| | 7.9.5 | Others | |
| 8. | R | EFERENCES | |
| | | | 15 |
| 10 | н | ISTORY TABLE | 16 |

## 1. LIST OF ABBREVIATIONS

| Term | Definition / description |
|--------|-----------------------------------------------|
| AE | Adverse event |
| ADR | Adverse Drug Reaction |
| ANOVA | Analysis of Variance |
| BMI | Body Mass Index |
| CRF | Case report form |
| CKD | Chronic Kidney Disease |
| DBLM | Database lock meeting |
| eGFR | Estimated Glomerular Filtration Rate |
| FAS | Full Analysis Set |
| HbA1c | Glycated Haemoglobin A1c |
| ICH | International Conference on Harmonisation |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NSP | Non-interventional Study Protocol |
| PT | Preferred term |
| PV | Protocol violation |
| Q1 | Lower quartile |
| Q3 | Upper quartile |
| RPM | Report planning meeting |
| SD | Standard deviation |
| SEAP | Statistical and Epidemiological Analysis Plan |
| SOC | System organ class |
| T2DM | Type 2 Diabetes Mellitus |

## 2. INTRODUCTION

As per International Conference on Harmonisation (ICH) guideline E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Statistical and Epidemiological Analysis Plan (SEAP) assumes familiarity with the Non-interventional Study Protocol (NSP). In particular, the SEAP is based on the planned analysis specification as written in NSP Section 9 "Research Methods". Therefore, SEAP readers may consult the NSP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size.

## 3. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

Three additional further outcomes (Hyperuricemia, Hypercholesteremia and Hypertriglyceridemia) are identified from the lab test results, and collected on eCRF, due to the consideration that missing values of lab tests results are inevitable and those diagnosis/diseases are more interested outcomes. In the analyses, they will be considered as part of medical history.

The analysis population Full Analysis Set (FAS), which includes all patients with an HbA1c measurement, is modified to: Full Analysis Set – Eligible (FAS – E), which includes all eligible patients regarding to inclusion and exclusion criteria with an HbA1c measurement.

Two additional sets, FAS – E with Hypoglycaemia and FAS – E with Hypoglycaemia leading to therapy change, are created for the analysis of treatment pattern.

## 5. OUTCOMES

#### 5.1 MAIN OUTCOMES

The primary outcome is the proportion of patients attaining blood glucose control target of HbA1c<7%.

NSP 9.3.2 defines the following parameters as secondary outcomes:

- Renal function level of patients
- Treatment regimens for T2DM that patient are currently taking
- Proportion of macro-vascular and micro-vascular diabetic complications
- Proportion of Hypoglycaemic occurrence
- Proportion of Hypoglycaemia leading to therapy change
- Proportion of Anti-hypertension therapy usage
- Proportion of Lipid Lowering therapy usage
- Proportion of Anti-Platelet therapy usage
- Treatment adherence to Chinese T2DM guideline 2013

#### 5.3 OTHER VARIABLES

All adverse drug reactions (ADRs) (serious and non-serious) and all AEs with fatal outcome (death) for any BI drug approved for the indication of T2DM must be collected by the investigator from signing the informed consent onwards until the end of the study.

#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 EXPOSURE

Not applicable.

#### 6.2 IMPORTANT PROTOCOL VIOLATIONS

Not applicable.

#### 6.3 PATIENT SETS ANALYSED

- Full Analysis Set Eligible (FAS E):
  The FAS E includes all eligible patients regarding to inclusion and exclusion criteria with an HbA1c measurement.
- FAS Albuminuria:

The FAS – Albuminuria dataset is a subset of patients of FAS – E, which includes T2DM patients with albuminuria (micro-albuminuria without urinary tract infection based on urine WBC result and macro-albuminuria).

- FAS E with Hypoglycaemia: The FAS – E with Hypoglycaemia dataset is a subset of patients of FAS – E, which includes T2DM patients with Hypoglycaemia as medical history.
- FAS E with Hypoglycaemia leading to therapy change: The FAS – E with Hypoglycaemia leading to therapy change dataset is a subset of patients of FAS – E, which includes T2DM patients with Hypoglycaemia leading to therapy change as medical history.

## 6.5 HANDLING OF MISSING DATA AND OUTLIERS

If patients have missing values for an outcome, those patients will be excluded for that outcome's analysis. No imputation approach will be applied. Any removal from the analysis will be documented.

# 6.6 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Not applicable.

## 7. PLANNED ANALYSIS

The following standard descriptive statistical parameters will be displayed in summary tables of all continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all subjects in the respective subject set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

For logistic regression model, adjusted odds ratio with 95% confidence interval, and p-value will be provided for the factors involved.

All data processing, summarization and analyses will be performed using Version 9.2 (or later) of the SAS statistical software package (Windows OS).

### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Summary statistics will be provided for the following demographics and baseline characteristics: Age, Age category, Gender, Education level, Smoking history, Physical activity, Body height, Body weight, BMI, Waist circumference, Heart rate, Systolic blood pressure, Diastolic blood pressure, Medical history, Treatment adherence to Chinese T2DM guideline 2013, Family history, Follow-up duration and Albuminuria. Descriptive statistics will be presented for continuous variables. Frequency and proportion will be used to summarize categorical variables. These will be based on both FAS – E and FAS – Albuminuria.

By-subject listings will be produced accordingly.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

The treatment pattern for T2DM will be summarized descriptively with frequency and proportion on FAS – E, FAS – E with Hypoglycaemia, FAS – E with Hypoglycaemia leading to therapy change, and FAS – Albuminuria.

The proportion of using anti-hypertension therapy, lipid-lowering therapy, and antiplatelet therapy will be calculated respectively. The concomitant medications will be coded according to the most recent version of the World Health Organization – Drug Dictionary

SEAP for BI Trial No: 1218.174 Page 11 of 16

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Enhanced/Herbal Dictionary (WHO DDE/HD), and summarized by ATC level 4 and preferred term.

The proportion of each macro-vascular and micro-vascular diabetic complication will be summarized respectively.

By-subject listings will be produced accordingly.

#### 7.3 METHODS ADDRESSING BIAS

Not applicable.

# 7.4 METHODS ADDRESSING CONFOUNDING / EFFECT MEASURE MODIFICATION

Identified confounders will be included in the logistic regression model to adjust the main outcome result. However unidentified confounders cannot be controlled for using statistical analyses.

#### 7.6 MAIN ANALYSES

The blood glucose control proportion (HbA1c<7%) will be tabulated on FAS – E.

The analyses for parameters below will be performed on both FAS – E and FAS – Albuminuria:

- Renal function variables (eGFR, albuminuria, and CKD staging) will be summarized
- The proportion of the occurrence of hypoglycaemia and the proportion of hypoglycaemia leading to therapy change will be summarized descriptively.

#### 7.8 EXPOSURE TIME

Not applicable.

#### 7.9 SAFETY ANALYSIS

#### 7.9.1 Adverse events

AEs will be summarized on both FAS – E and FAS – Albuminuria.

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs.

An overall summary of adverse events will be presented.

Adverse events will be coded according to the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA). The frequency of subjects with adverse events will be summarized by treatment, system organ class and preferred term. The system organ classes will be sorted in alphabet order, preferred terms will be sorted by frequency (within system organ class).

#### 7.9.2 Laboratory data

Refer to section 7.7 of this document.

#### 7.9.3 Vital signs

Refer to section 7.1 of this document.

#### 7.9.4 ECG

Not applicable.

#### **7.9.5** Others

The subject disposition summaries will be provided. The number of enrolled subjects and of entered subjects will be included. The completion status of data collection and the reason for discontinuation will be summarized.

By-subject listing will be provided.

# 8. REFERENCES

1 001-MCS-50-413\_RD-01: "Protocol Violation Handling Definitions", current version, IDEA for CON.

# 10. HISTORY TABLE

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| No. | (dd Mmm yyyy) | | changed | |
| 1.0 | 09Feb2018 | | NA | Final version before database lock. |